CLINICAL TRIAL: NCT07325110
Title: Interoceptive Awareness and Function in Adolescents With Chronic Pain
Status: Recruiting | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 25-077
Record Dates: First submitted 2025-11-11; First posted 2026-01-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Chronic Pain Syndrome; Pain, Chronic
Keywords: chronic pain; adolescents; interoceptive awareness; function; occupational therapy; yoga
MeSH Terms: conditions — Chronic Pain | interventions — Occupational Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Participants who are diagnosed with a form of chronic pain and are referred for occupational therapy treatment services.
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Other: Occupational Therapy — Participants will receive an occupational therapy treatment plan of care that includes yoga for 8-12 weekly visits. They will complete pre and post questionnaires to measure their interoceptive awareness and function.

SUMMARY:
The main objectives of this study are to compare the levels of interoceptive awareness and self-reported function pre and post completion of an occupational therapy treatment plan. The target population are adolescents aged 11-21 years that are diagnosed with chronic pain and are seen through the Pain Team at Connecticut Children's. The primary aims are:

* To compare the reported levels of interoceptive awareness in adolescents with chronic pain before and after their occupational therapy treatment plan.
* To compare the reported levels of function in adolescents with chronic pain before and after their occupational therapy treatment plan.

DETAILED DESCRIPTION:
Background:

There has been an increasing number of adolescents with chronic pain who have been referred to pain team and to occupational therapy (OT) for intervention. The investigators on this study have been using the multifaceted intervention of yoga to treat this complex impairment. The main objectives of this study are to compare the level of interoceptive awareness and self-reported function pre and post completion of an occupational therapy treatment plan. The target population are adolescents, aged 11-21 years, that are diagnosed with chronic pain and are seen through the pain team at Connecticut Children's. Data will be collected pre and post occupational therapy treatment plan through use of the Multidimensional Assessment of Interoceptive Awareness (MAIA) to look at possible changes in interoception and the Patient-Reported Outcomes Measurement Information System (PROMIS) to look at possible changes in function. Interoception is the 8th sensory system or the sense of internal bodily signals and interoceptive awareness is the ability to be aware of and respond to these sensations. The areas of function on the PROMIS are Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Peer Relationships/Social Roles and Activities, and Pain Interference. These participants will also complete a 4 question 3 month follow up survey. The participants in the study are a convenience sample of patients referred to therapy services from Pain Team visit.

Study Procedures:

Study Participants

1. Consent/assent will take place at the pain team visit within a private treatment room by one of the study team members. The participant and family will be given a detailed description of the purpose of the study and expectations for participants. The participant and family will have the opportunity to read the consent forms and ask any questions the participant and/or family may have about the research.
2. If the participant agrees to enroll in the study, the participant will be asked to complete the electronic signature in Research Electronic Data Capture (REDCap) to complete the consenting process. A paper version will be available if needed.
3. If in the scenario where a legal guardian is not present and required for consent, remote consenting will be offered to fulfill consenting requirements. A copy will be provided upon completion.
4. All patients that are seen by the pain team and referred to the occupational therapy department at Connecticut Children's and consent for this study will begin therapy services within one month of being seen in clinic.
5. During the first visit, the PROMIS and MAIA pre-test will be provided to the participant for completion within REDCap. A paper version will be available if needed and then inputted into REDCap by investigator.
6. Over the twelve sessions, participants will be educated on and complete components of breathwork, mindfulness, and poses. These will be individualized for each participant, based on the participant's abilities and needs, from a list that has been developed along with a general outline of the progression of sessions.
7. At the end of each session, a home program will be provided based off of concepts learned in treatment with expectation of implementation 3x per week.
8. At the start of each visit, attendance will be recorded into REDCap and the participant will report the number of home program sessions completed since last visit and will be recorded in REDCap.
9. During the last visit, the PROMIS and MAIA post-test will be provided to the participant for completion within REDCap. A paper version will be available if needed and then inputted into REDCap by investigator.
10. A 3 month follow-up survey will be sent via email to all participants in the research group.

Data Collection and Management:

Allison Fell OTR/L and Samantha DeFrancesco OTR/L will oversee data management.

1. Data collection forms: All data points and outcome measures will be completed and entered into a REDCap database to secure data and facilitate data analysis.
2. Data collection software: The Research Operations and Development team assisted with the development of this REDCap project. The data will be collected by investigators, and it will be stored only in REDCap. The database will only be accessible to those individuals included in this study.
3. Patient demographic data will be entered into REDCap- this would include the Medical Record Number (MRN), Date of birth, Sex/Gender, Race/ethnicity, Diagnosis, Insurance type, Email, and Phone number to allow for improved ease and accuracy of data collection. All other clinical data will be stored in REDCap. The data will be collected by investigators, and it will be entered into REDCap by Allison Fell OTR/L and Samantha DeFrancesco OTR/L to ensure data accuracy.
4. Once data have been reviewed as stated above, medical record numbers will be removed from the main dataset. A separate file will be kept to link patient names and identification and medical record numbers. This will be used to keep a list of patients in case charts need to be re-visited to collect additional data.
5. Record retention and confidentiality will be dictated by the current procedures at Connecticut Children's. All information will be stored in a password protected database and on a password protected computer. No access to information is possible from an outside source.

Patient confidentiality statement:

Strict measures will be required for respecting and maintaining patient confidentiality. Collection of a patient identifier including medical record numbers and the patients name is necessary to ensure comprehensive inclusion of eligible subjects and accurate linking of data from different data sets. The database used for the study will be password protected and stored in REDCap. Once the study investigators have collected all the data, the data set will be frozen for analysis. At this time, the study investigators will completely de-identify all subjects. Medical record numbers as well as the patient's names will be removed and patients will be referred to by study number only. De-identification will take place once the study investigators have collected all data. The study investigators expect that these measures will minimize any risk to confidentiality very effectively, and that any unavoidable residual risk will be balanced generously by the potential benefit to society of the knowledge that will be obtained through this research.

Sample Size Justification:

For participant change the investigators will need 34 OT completers to provide ≥80% power for 0.5 Standard Deviation (SD) improvement.

Feasibility, Accrual, and Expected Duration of Accrual:

Over 200 new patients were referred to pain team last year in 2024. The study investigators plan to recruit as many of these patients that meet criteria to achieve a medium effect sample size within a 12-month duration.

Study Limitations:

There are several limitations anticipated with this study. These limitations include a small sample size from a single institution, no control group, and potential bias with patient selection.

Use of Study Results:

The outcomes of this study will be used to assist in quality improvement within the department and guide future research questions. The investigators plan to publish results in a peer-reviewed publication and to present the findings at a conference.

ELIGIBILITY:
Study Group:

Inclusion Criteria:

1. Adolescents seen as new patients in the pain clinic at Connecticut Children's
2. Referred to occupational therapy services.
3. Adolescents diagnosed with a form of chronic pain.
4. Between the ages of 11 and 21 years at time of enrollment.
5. If over 18, the ability to understand and willingness to sign the informed consent document or the ability to use the short form process.
6. If under 18, the parent/legal guardian, has the ability to understand and willingness to sign the informed consent document or the ability to use the short form process.
7. Adolescents between the ages of 11 and less than 18 years with the ability to understand and willingness to sign assent.
8. Adolescents who agree to therapeutic yoga as a planned part of their occupational therapy treatment plan.

Exclusion Criteria:

1. Adolescents not receiving yoga as an element of their occupational therapy treatment plan.
2. Adolescents with a cognitive impairment that would impede their ability to participate.
3. Adolescents with a neuromuscular diagnosis, such as Cerebral Palsy, Spinal Muscular Atrophy, and Muscular Dystrophies, that are not appropriate for yoga as an element of their treatment plan for this study.
4. Adolescents unwilling to complete surveys to participate in this research study.
5. Adolescents who are currently actively practicing yoga
6. Adolescents who are currently receiving occupational therapy at another location.

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants for this study are patients seen within the Pain Team Clinic at Connecticut Children's. They are adolescents aged 11-21 years old that are diagnosed with a form of chronic pain and are referred for occupational therapy services.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Profile GenPop v.3 | Assessment administered at the first therapy treatment visit and last treatment visit within a 4 month time frame.
  For ages 8-17. The PROMIS is a system that measures how patients feel and function in terms of their physical, mental, and social health. It measures pain, fatigue, physical functioning, emotional distress, and social role participation. PROMIS uses a series of questions to assess how patients feel and what they are able to do. It is a total of 36 questions with a collection of 5- and 6-item short forms assessing anxiety, depressive symptoms, fatigue, pain interference, physical function-mobility, and peer relationships, as well as a single pain intensity item. For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation (SD) of 10 because calibration testing was performed on a large sample of the general population. The T-score is provided with an error term. A higher PROMIS T-score represents more of the concept being measured. A PROMIS score includes a T-score and a standard error (SE).
Patient-Reported Outcomes Measurement Information System (PROMIS)-43 Profile v2.1 | Assessment administered at the first therapy treatment visit and last treatment visit within a 4 month time frame.
  For ages 18+. The PROMIS is a system that measures how patients feel and function in terms of their physical, mental, and social health. It measures pain, fatigue, physical functioning, emotional distress, and social role participation. PROMIS uses a series of questions to assess how patients feel and what they are able to do. It is a total of 43 questions with a collection of 6-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item. For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation (SD) of 10 because calibration testing was performed on a large sample of the general population. The T-score is provided with an error term. A higher PROMIS T-score represents more of the concept being measured. A PROMIS score includes a T-score and a standard error (SE).
Multidimensional Assessment of Interoceptive Awareness- Version 2 | Assessment administered at the first therapy treatment visit and last treatment visit within a 4 month time frame.
  For ages 18+. The Multidimensional Assessment of Interoceptive Awareness is a patient reported questionnaire with 37-items to measure multiple dimensions of interoception (body awareness) through an 8-subscale state-trait questionnaire. The areas this assessment measures are noticing, non-distracting, not worrying, attention regulation, emotional awareness, self-regulation, body listening, and trust.
  Scoring: Scores are between 0 and 5, where higher score equates to more awareness of bodily sensation. A percentile is also calculated, indicating how the responded scored in comparison to a normative sample. Interpretation using percentiles helps contextualize scores. For example, percentile below 50 indicate that the individual scored below what is typical. Extreme percentile scores (below 10 or above 90) are of particular clinical significance.
Multidimensional Assessment of Interoceptive Awareness- Youth | Assessment administered at the first therapy treatment visit and last treatment visit within a 4 month time frame.
  For ages 7-17. The Multidimensional Assessment of Interoceptive Awareness is a patient reported questionnaire with 32-items to measure multiple dimensions of interoception (body awareness) through an 8-scale state-trait questionnaire. The areas this assessment measures are noticing, non-distracting, not worrying, attention regulation, emotional awareness, self-regulation, body listening, and trust.
  Scoring: Scores are between 0 and 5, where higher score equates to more awareness of bodily sensation. A percentile is also calculated, indicating how the responded scored in comparison to a normative sample. Interpretation using percentiles helps contextualize scores. For example, percentile below 50 indicate that the individual scored below what is typical. Extreme percentile scores (below 10 or above 90) are of particular clinical significance.

SECONDARY OUTCOMES:
3 Month Follow-up Survey | Survey will be sent out to study group participants 3 months after their last occupational therapy treatment visit.
  4 question survey to assess participant continued use of strategies learned in therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Fell, BS, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chambers CT, Dol J, Tutelman PR, Langley CL, Parker JA, Cormier BT, Macfarlane GJ, Jones GT, Chapman D, Proudfoot N, Grant A, Marianayagam J. The prevalence of chronic pain in children and adolescents: a systematic review update and meta-analysis. Pain. 2024 Oct 1;165(10):2215-2234. doi: 10.1097/j.pain.0000000000003267. Epub 2024 May 15. PMID 38743558
- [Background] Craig AD. How do you feel--now? The anterior insula and human awareness. Nat Rev Neurosci. 2009 Jan;10(1):59-70. doi: 10.1038/nrn2555. PMID 19096369
- [Background] Eccleston C, Malleson P. Managing chronic pain in children and adolescents. We need to address the embarrassing lack of data for this common problem. BMJ. 2003 Jun 28;326(7404):1408-9. doi: 10.1136/bmj.326.7404.1408. No abstract available. PMID 12829527
- [Background] Evans S, Moieni M, Sternlieb B, Tsao JC, Zeltzer LK. Yoga for youth in pain: the UCLA pediatric pain program model. Holist Nurs Pract. 2012 Sep-Oct;26(5):262-71. doi: 10.1097/HNP.0b013e318263f2ed. PMID 22864296
- [Background] Gnall KE, Sinnott SM, Laumann LE, Park CL, David A, Emrich M. Changes in Interoception in Mind-body Therapies for Chronic Pain: A Systematic Review and Meta-Analysis. Int J Behav Med. 2024 Dec;31(6):833-847. doi: 10.1007/s12529-023-10249-z. Epub 2024 Jan 2. PMID 38169051
- [Background] Hechler T. Altered interoception and its role for the co-occurrence of chronic primary pain and mental health problems in children. Pain. 2021 Mar 1;162(3):665-671. doi: 10.1097/j.pain.0000000000002099. No abstract available. PMID 33021565
- [Background] Horsburgh A, Summers SJ, Lewis A, Keegan RJ, Flood A. The Relationship Between Pain and Interoception: A Systematic Review and Meta-Analysis. J Pain. 2024 Jul;25(7):104476. doi: 10.1016/j.jpain.2024.01.341. Epub 2024 Jan 18. PMID 38244898
- [Background] Kempert H. The Use of Yoga as a Group Intervention for Pediatric Chronic Pain Rehabilitation: Exploring Qualitative and Quantitative Outcomes. Int J Yoga. 2020 Jan-Apr;13(1):55-61. doi: 10.4103/ijoy.IJOY_13_19. PMID 32030022
- [Background] Khalsa SS, Adolphs R, Cameron OG, Critchley HD, Davenport PW, Feinstein JS, Feusner JD, Garfinkel SN, Lane RD, Mehling WE, Meuret AE, Nemeroff CB, Oppenheimer S, Petzschner FH, Pollatos O, Rhudy JL, Schramm LP, Simmons WK, Stein MB, Stephan KE, Van den Bergh O, Van Diest I, von Leupoldt A, Paulus MP; Interoception Summit 2016 participants. Interoception and Mental Health: A Roadmap. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):501-513. doi: 10.1016/j.bpsc.2017.12.004. Epub 2017 Dec 28. PMID 29884281
- [Background] Khalsa SB, Butzer B. Yoga in school settings: a research review. Ann N Y Acad Sci. 2016 Jun;1373(1):45-55. doi: 10.1111/nyas.13025. Epub 2016 Feb 25. PMID 26919395
- [Background] Koechlin H, Donado C, Locher C, Kossowsky J, Lionetti F, Pluess M. Sensory processing sensitivity in adolescents reporting chronic pain: an exploratory study. Pain Rep. 2023 Jan 6;8(1):e1053. doi: 10.1097/PR9.0000000000001053. eCollection 2023 Jan. PMID 36699990
- [Background] Lucas JW, Sohi I. Chronic Pain and High-impact Chronic Pain in U.S. Adults, 2023. NCHS Data Brief. 2024 Oct;(518):CS355235. doi: 10.15620/cdc/169630. PMID 39751180
- [Background] Mehling W. Differentiating attention styles and regulatory aspects of self-reported interoceptive sensibility. Philos Trans R Soc Lond B Biol Sci. 2016 Nov 19;371(1708):20160013. doi: 10.1098/rstb.2016.0013. Epub 2016 Oct 10. PMID 28080970
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Background] Salaffi F, Sarzi-Puttini P, Atzeni F. How to measure chronic pain: New concepts. Best Pract Res Clin Rheumatol. 2015 Feb;29(1):164-86. doi: 10.1016/j.berh.2015.04.023. Epub 2015 Jun 19. PMID 26267010